CLINICAL TRIAL: NCT00785876
Title: Controlled Radiography for Ankle Injury Cases in Kids in the Emergency Department: Implementation of the Low Risk Ankle Rule
Brief Title: Implementation of the Low Risk Ankle Rule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Kathy Boutis, Staff Physician, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000012792
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Ankle Injury
Keywords: Paediatric; Emergency Department; Ankle; Injury; Low risk ankle rule
MeSH Terms: conditions — Ankle Injuries; Emergencies; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Control Sites
- 2 (Experimental): Intervention Sites
  Interventions: Other: LRAR Implementation

INTERVENTIONS:
Other: LRAR Implementation — Pre-LRAR - no changes in the usual procedures for the first 26 weeks except for flagging of all paediatric charts with ankle injuries, ED documentation which will not refer to the LRAR and phone follow up.
  Post-LRAR: At 27 weeks, in addition to the aforementioned ED collection sheet and phone follow up, the implementation strategy for the LRAR rule and related management will be introduced at the intervention hospitals.
  Arms: 2

SUMMARY:
Ankle injuries are a very common injury in children. Each year approximately 35000 kids present to Ontario emergency departments (ED) with this problem. Right now, about 90% of these children get x-rays of the injured ankle, even though only 12% of these x-rays show a break in the bone. Some excellent research has created some rules that doctors can use to help them decide which children really need x-rays. Unfortunately, even though these rules have been proven to safely reduce x-rays by as much as two-thirds, most doctors are not using these rules.

Therefore, this study will be the first to put the best paediatric ankle x-ray rule, the Low Rick Ankle Rule, into physician practice in EDs. Our main goal is to determine how much we can reduce ankle x-ray rates in EDs that use this rule regularly versus those that do not. If we show that doctors can safely use this rule regularly and the number of ankle x-rays will be significantly less, this will lessen unnecessary potentially harmful radiation exposure in children, these children will spend less time in an ED, and the health care system will save money.

ELIGIBILITY:
Inclusion Criteria:

* All otherwise healthy children between the ages of 3 and 16 years of age that present to the participating EDs with an isolated acute (< 72 hours) blunt ankle injury due to any mechanism of injury will be eligible for the study. The age criteria were chosen to match those ages in which the LRAR was validated.

Exclusion Criteria:

1. Children with ankle injuries who were referred from outside the hospital with radiographs.
2. Children with ankle injuries who returned for reassessment of the same ankle injury.
3. Children with open wounds on their ankle and/or foot
4. All children at risk for pathological fractures such as those with congenital or acquired generalized bony disease (Appendix I). Clinical presentation and risks in these cases may be altered.
5. Congenital anomalies of the feet and/or ankles (eg club feet, tarsal coalition). These abnormalities may have features which may complicate clinical assessment.
6. Patients with known coagulopathies. Underlying hemarthrosis may complicate clinical assessment.
7. Patients with cognitive and/or developmental delay. These patients may not localize pain.
8. Injuries greater than 72 hours old. The signs and symptoms of the most common fracture, the Salter-Harris I fracture of the distal fibula, may be diminished. Our ability to make this clinical diagnosis with confidence may thus be compromised.
9. Recent history of surgery or closed reduction of the same ankle within the last 3 months. These prior events may confuse current presenting symptomatology and ability to weight-bear and recover normally.
10. Patients with low risk injuries who do not have phone or electronic mail access and/or have an insurmountable language barrier. This will preclude follow up.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To assess the impact of a LRAR implementation strategy on paediatric ankle radiography rates in participating EDS. | three six month phases of implementation

SECONDARY OUTCOMES:
Ankle x-ray rate changes at individual hospital from pre-LRAR to post-LRAR implementation phases. | duration of subjects participation in study
Intervention and control sites will be compared individually and collectively, during the post-LRAR for: missed significant fractures, number of unscheduled x-rays following initial ED visit, total length of stay, patient and physician satisfaction | duration of subjects participation in study
To determine the sustainability of the clinical impact of the LRAR strategy at intervention sites by comparing high and low intensity implementation phases with respect to weekly x-ray rates, missed fractures and physician and patient satisfaction | duration of subjects participation in study
To evaluate the performance of the LRAR during the implementation period of the rule at intervention sites with respect to: sensitivity and specificity of the LRAR for detecting "high risk" fractures and physician compliance with use of the rule | duration of subjects participation in study
To compare total costs of "low risk injuries" at intervention versus control sites during the post-LRAR implementation phase. | duration of subjects participation in study

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Boutis, MD, Principal Investigator — The Hospital for Sick Children
Locations (4):
- Canada (4):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Toronto East General Hospital, Toronto, Ontario

REFERENCES:
- [Result] Boutis K, Grootendorst P, Willan A, Plint AC, Babyn P, Brison RJ, Sayal A, Parker M, Mamen N, Schuh S, Grimshaw J, Johnson D, Narayanan U. Effect of the Low Risk Ankle Rule on the frequency of radiography in children with ankle injuries. CMAJ. 2013 Oct 15;185(15):E731-8. doi: 10.1503/cmaj.122050. Epub 2013 Aug 12. PMID 23939215
- [Result] Boutis K, von Keyserlingk C, Willan A, Narayanan UG, Brison R, Grootendorst P, Plint AC, Parker M, Goeree R. Cost Consequence Analysis of Implementing the Low Risk Ankle Rule in Emergency Departments. Ann Emerg Med. 2015 Nov;66(5):455-463.e4. doi: 10.1016/j.annemergmed.2015.05.027. Epub 2015 Jul 14. PMID 26187612
- See also: Link to Abstract: : Ann Emerg Med. 2015 Nov;66(5):455- — https://www.ncbi.nlm.nih.gov/pubmed/26187612
- See also: Link to Abstract: Effect of the Low Risk Ankle Rule on the frequency of radiography in children with ankle injuries. — https://www.ncbi.nlm.nih.gov/pubmed/23939215